CLINICAL TRIAL: NCT05435638
Title: Phase I, Open Label Study Designed to Evaluate the Safety and Efficacy of a 1% Topical Formulation of KM-001 in the Treatment of Type I Punctate Palmoplantar Keratoderma or Pachyonychia Congenital Diseases
Brief Title: Study Designed to Evaluate Safety and Efficacy of 1% Topical Formulation of KM-001 on Type 1 Punctate Palmoplantar Keratoderma or Pachyonychia Congenita Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kamari Pharma Ltd (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KM-001B1
Record Dates: First submitted 2022-05-11; First posted 2022-06-28 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Punctate Palmoplantar Keratoderma Type 1; Pachyonychia Congenita
MeSH Terms: conditions — Keratosis palmoplantaris papulosa; Pachyonychia Congenita | interventions — Hematologic Tests; Urinalysis; Physical Examination; Vital Signs; Therapeutics; Pain Measurement; KPNA1 protein, human

STUDY DESIGN:
Intervention Model Description: Patients with type I punctate palmoplantar keratoderma or pachyonychia congenita will be recruited to be treated, with 1% topical KM-001.
  Arm 1: up to 10 eligible patients will be treated twice daily for 12 weeks. Treatment safety and efficacy will be assessed in the clinic visits up to day 84. In between, safety will also be assessed by phone. PK blood samples will be collected. 1 week after the end of treatment visit, patients will return to the clinic for final safety, efficacy and PK evaluations.
  Arm 2: up to 8 eligible patients, will be treated twice daily, for 16 weeks, with 1% topical KM-001. Treatment safety and efficacy will be assessed in the clinic visits up to day 112. PK blood samples will be collected. In between visits, safety will also be assessed by phone. 2 weeks after the end of treatment visit, patients will return to the clinic for final safety, efficacy, and PK evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KM-001 1% cream 12 weeks treatment (Experimental): KM-001 1% cream will be applied to the affected area, twice daily for 12 consecutive weeks.
  KM-001 will be supplied in glass jars (30 g) and will be provided to patients with spatulas and polyethylene gloves.
  Interventions: Diagnostic Test: Serum chemistry; Diagnostic Test: Hematology; Diagnostic Test: Urinalysis; Diagnostic Test: Physical Examination; Diagnostic Test: Vital Signs; Diagnostic Test: ECG Test; Diagnostic Test: PK; Diagnostic Test: IGA scoring; Drug: KM-001 1% cream 12 weeks treatment; Diagnostic Test: Clinician global impression of severity (CGI-S); Diagnostic Test: Visual Analogue Scale (VAS); Diagnostic Test: Patient global impression of change (PGI-C) scoring; Diagnostic Test: Patient global impression of severity (PGI-S) scoring; Diagnostic Test: Lesion photography
- KM-001 1% cream 16 weeks treatment (Experimental): KM-001 1% cream will be applied to the affected area, twice daily for 16 consecutive weeks.
  KM-001 will be supplied in glass jars (30 g) and will be provided to patients with spatulas and polyethylene gloves.
  Interventions: Diagnostic Test: Serum chemistry; Diagnostic Test: Hematology; Diagnostic Test: Urinalysis; Diagnostic Test: Physical Examination; Diagnostic Test: Vital Signs; Diagnostic Test: ECG Test; Diagnostic Test: PK; Diagnostic Test: IGA scoring; Diagnostic Test: Clinician global impression of severity (CGI-S); Diagnostic Test: Visual Analogue Scale (VAS); Diagnostic Test: Patient global impression of change (PGI-C) scoring; Diagnostic Test: Patient global impression of severity (PGI-S) scoring; Diagnostic Test: Lesion photography; Drug: KM-001 1% cream 16 weeks treatment

INTERVENTIONS:
Diagnostic Test: Serum chemistry — Approximately 5 mL whole blood will be collected after an ≥8 h fast for complete blood count (CBC) during Screening, and on Days 7 and 84 of treatment, at early termination (ET), if required, and at the EoT (Arm 2: Day 112) and follow-up EoS visits (Cohort 1: Day 91; Cohort 2: Day 126).
  Serum chemistries will include assessment of total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), lactate dehydrogenase (LDH), alkaline phosphatase, glucose, sodium, potassium, blood urea nitrogen (BUN), and creatinine.
Diagnostic Test: Hematology — Approximately 5 mL whole blood will be collected after an ≥8 h fast for complete blood count (CBC) during Screening, and on Days 7 and 84 of treatment, at early termination (ET), if required, and at the EoT (Arm 2: Day 112) and follow-up EoS visits (Cohort 1: Day 91; Cohort 2: Day 126). The CBC assessment will include a red blood cells (RBC), hemoglobin, hematocrit, platelet count, mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), mean platelet volume (MCV), white blood cells (WBC), neutrophils (% and abs.), lymphocytes (% and abs.), monocytes (% and abs.), eosinophils (% and abs.), basophils (% and abs.), large unstained cells (% and abs.).
Diagnostic Test: Urinalysis — General urinalysis will be performed, by dipstick, during Screening, on Days 7 and 84 of treatment, at early termination (ET), if required, and at the EoT (Cohort 2: Day 112) and follow-up EoS visits (arm 1: Day 91; Arm 2: Day 126).
  Approximately 7-10 mL urine will be collected. Urinalysis will include pH, specific gravity, blood, nitrites, glucose, ketones, protein, bilirubin urobilinogen and leukocytes. A microscopic examination of the urine will be performed only if clinically indicated.
Diagnostic Test: Physical Examination — A complete physical examination will be performed at Screening, at all in-clinic study visits, and at the End of Study visit.
  The physical examination will cover a careful assessment of all body systems, including the head, eyes, ears, nose, and throat and the respiratory, cardiovascular, GI, urogenital, musculoskeletal, neurological, dermatological, hematologic/lymphatic, and endocrine systems. Particular attention will be placed on the areas affected by the disease.
  • Symptom-directed physical examinations will be performed at all other study visits.
Diagnostic Test: Vital Signs — Vital sign measurements (body temperature, pulse and resting systolic and diastolic blood pressure) will be measured at Screening, at all in-clinic study visits, and at the End of Study visit. Vital signs will be measured in supine position after at least five minutes of rest.
Diagnostic Test: ECG Test — A 12-lead, resting, digital ECG will be taken for each participant during Screening, on Days 42 and 84 (for both arms), and on day 112 (Arm 2 only), after the patient has been supine for at least 5 min. At minimum, the following ECG parameters will be recorded: heart rate (HR), PR, QT and QRS intervals and QTC. The report will be signed by the Investigator, who will record in the CRF whether it is normal, abnormal but not clinically significant, or abnormal AND clinically significant. In the latter case the eligibility of the participants will be reviewed.
Diagnostic Test: PK — Blood PK analyses will be performed on ≥5ml blood collected in 5-mL K-EDTA CRO coded pre-labeled tubes, refrigerated immediately after collection. Plasma will be separated by centrifugation within 2h, and then frozen at -20C.
  Blood samples will be collected pre-dose on Days 0, 7, and 84, as well as pre-dose at EoT (Arm 2: Day 112), and at any point during the in-clinic visit at EoS (Arm 1: Day 91; Arm 2: Day 126).
Diagnostic Test: IGA scoring — Lesions severity will be assessed using the Investigator's Global Assessment (IGA) scale,which is a 5-point scale (from 0 ="no disease" to 4="severe disease") based on Simpson et al. 2020, IGA for atopic dermatitis (see Table 4; Simpson et al. 2020).
  The IGA score is selected using the descriptors below that best describe the overall appearance of the lesions at a given timepoint. It is not necessary that all characteristics under morphological description are present. Excoriations should not be considered when assessing disease severity.
Drug: KM-001 1% cream 12 weeks treatment — KM-001 1% cream will be applied to the treated area twice daily for 12 consecutive weeks, 2 gr per treatment, and overall, 4 gr of daily dose.
  KM-001 will be supplied in glass jars (30 g) and will be provided to patients with spatulas and polyethylene gloves.
  Other Names: Cohort 1
  Arms: KM-001 1% cream 12 weeks treatment
Diagnostic Test: Clinician global impression of severity (CGI-S) — Lesions severity will be assessed using the CGI-S scale, which is a 5-point scale (from 0= "none" to 4= "very severe") modified from Busner et al. 2007 (30) by the investigator at screening and on Days 0, 7, 28, 42, 63, 84, 91, 112, and 126 (as applicable, per arm), and at ET visit, if applicable.
  The clinician scoring takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms (pain), behaviour, and the impact of the symptoms on the patient's ability to function (ability to walk). investigators will complete the CGI-S at various timepoints based on the question. "Please choose the response that best describes your assessment of the disease severity, based upon the totality of information available to you"
Diagnostic Test: Visual Analogue Scale (VAS) — The VAS score will be collected on every in-clinic visit during the treatment period (Days 0, 7, 28, 42, 63, 84, 91, 112, and 126 (as applicable, per arm), and at ET visit, if applicable.).
  The PGIs will be evaluated on Days 0, 7, 28, 42, 63, 84, 91, 112, and 126 (as applicable, per arm), and
  The following parameter will be evaluated on a VAS from 0 (no pain) to 100 (severe intolerable pain) based on the question:
  "How was your worst pain intensity in the past 24 hours?"
Diagnostic Test: Patient global impression of change (PGI-C) scoring — The PGI-C scale was developed to provide a brief, stand-alone assessment of the patient's view of his/her global functioning prior to and after initiating a trial medication.
  The PGIs will be evaluated on Days 7, 28, 42, 63, 84, 91, 112, and 126 (as applicable, per arm), and at ET visit, if applicable.
  The PGI-C will be evaluated using a 7-point scale from 1 (very much improved) to 7 (very much worse) answering the question Since the start of the trial, my overall status has.
Diagnostic Test: Patient global impression of severity (PGI-S) scoring — The PGI-S scale was developed to provide a brief, stand-alone assessment of the patient's view of his/her global functioning prior to and after initiating a trial medication.
  The PGIs will be evaluated on Days 0, 7, 28, 42, 63, 84, 91, 112, and 126 (as applicable, per arm), and at ET visit, if applicable.
  The PGI-S will be evaluated using a 5-point scale from 1 (none) to 5 (very severe) answering the question Please rate the severity of your disease right now.
Diagnostic Test: Lesion photography — High-quality photographic documentation of the treated lesions will be performed on screening, and on Days 0, 7, 28, 42, 63, 84, 91, 112, and 126 (as applicable, per arm), and at ET visit, pre-dose, if applicable.
Drug: KM-001 1% cream 16 weeks treatment — KM-001 1% cream will be applied to the treated area twice daily for 12 consecutive weeks, 2 gr per treatment, and overall, 4 gr of daily dose.
  KM-001 will be supplied in glass jars (30 g) and will be provided to patients with spatulas and polyethylene gloves.
  Other Names: Cohort 2
  Arms: KM-001 1% cream 16 weeks treatment

SUMMARY:
In this phase 1 open label study for patients with type I punctate palmoplantar keratoderma or pachyonychia congenital, 2 arms will be recruited to be treated twice daily, with 1% topical KM-001.

Arm 1: up to 10 eligible patients will be treated for 12 weeks. Arm 2: up to 8 eligible patients will be treated for 16 weeks.

Treatment safety and efficacy will be assessed in the clinic visits (for arm 1 up to day 91, for arm 2 up to day 126). In between safety will also be assessed by phone visits.

At the in-clinic visits, treatment efficacy (lesion clearance - IGA, CGI-S, PGI-C, PGI-S and VAS pain) will also be assessed.

PK blood samples will be collected for arm 1: on Days 0, 7, 84 (EoT visit). One week after the end of treatment (EoT) visit, patients will return to the clinic for final safety, efficacy and PK evaluations. For arm 2, PK blood samples will be collected on days 0, 7, 84, 112 (EoT visit). Two weeks after the end of treatment (EoT) visit, patients will return to the clinic for final safety, efficacy and PK evaluations.

DETAILED DESCRIPTION:
The palmoplantar keratoderma (PPK) group of skin disorders results from various mutations in several epidermal genes and is characterized by thickening of the skin on the palms and soles.

Punctate palmoplantar keratoderma (PPKP1) is a rare autosomal, dominant, inherited skin disease characterized by bilateral asymptomatic, tiny, hyperkeratotic punctate papules and plaques on the palmoplantar surface.

Pachyonychia congenita (PC) is a rare group of autosomal dominant skin disorders that are caused by a mutation in one of five different keratin genes. PC is often associated with thickened toenails, plantar keratoderma, and plantar pain. Its manifestations include bilateral PPK on palms and soles pattern with sharp margins and a yellow tone.

A common characteristic of these skin diseases is the impaired differentiation of keratinocytes, often caused by defective calcium homeostasis. Normal calcium homeostasis is regulated by calcium ion channels, including the transient receptor potential cation channel subfamily V, member 3 (TRPV3), which has been implicated in regulation of keratinocyte proliferation, differentiation, and apoptosis. As a result, it has been suggested as a drug target for a variety of dermatological conditions and itch. It has therefore been suggested that inhibition of TRPV3 by specific antagonists can address the above-mentioned conditions.KM-001, developed by Kamari Pharma, is a potent and selective TRPV3 antagonist. Kamari has demonstrated that KM-001 reduces Ca+2flux in keratinocytes and decreases cell proliferation accompanied by normalization of keratinocyte differentiation markers. Efficacy was demonstrated in in vivo studies, using the DS-Nh mice model, where it was able to normalize epidermal hyperkeratosis. In addition, the compound significantly reduced pruritus which is characteristic of this model and of many types of PPK.

KM-001 topical formulation demonstrates favorable safety profile in rodents and minipigs and significant efficacy in animal models.

ELIGIBILITY:
Inclusion Criteria:

1. Read, understood and signed an informed consent form (ICF) before any investigational procedure(s) are performed.
2. Male or female and aged 18 - 75 years at the time of screening
3. Clinical diagnosis of:

   punctate keratoderma type I disease with confirmed heterozygous mutation in AAGAB gene OR pachyonychia congenita with confirmed heterozygous mutation in either KRT16, KRT17, KRT6A, KRT6B or KRT6C mutations.
4. The target treatment region is 0.5%-4% body surface area (BSA) including target lesions
5. CGI-S score of ≥2 (as assessed by the PI at screening).
6. Female patients of childbearing potential must agree to use a highly effective and approved method of contraception throughout the study and for 4 weeks after the last study drug administration. Male patients: female partners of male patients must use a reliable method of contraception during this study, and for 12 weeks after the last dose of study medications.
7. Female patients must refrain from donating eggs throughout the study and for 4 weeks after the last study drug administration. Male patients must refrain from sperm donation throughout the study and for 12 weeks after the last study drug administration.
8. Female patients of non-childbearing potential must meet one of the following criteria:

   * Absence of menstrual bleeding for 1 year prior to screening without any other medical reason.
   * Documented hysterectomy or bilateral oophorectomy at least 3 months before the study.
9. Patient is willing and able to comply with all time commitments and procedural requirements of the clinical study protocol.

Exclusion Criteria:

1. Known hypersensitivity or any suspected cross-allergy to the active pharmaceutical ingredient and/or excipients.
2. Regular alcohol consumption for males >21 units per week and for females >14 units per week (1 unit = 8gr of alcohol; e.g., 200 mL of 5% beer, 25 mL of 40% spirits or 125 mL of 8% wine).
3. Any medical or active psychological condition or any clinically relevant laboratory abnormalities, such as, but not limited, to elevated ALT or AST (>3 × upper limit of normal [ULN]) in combination with elevated bilirubin (>2 × ULN), at screening/ baseline that may put the patient at significant risk according to the investigator's judgment, if he/she participates in the clinical study, or may interfere with study assessments (e.g., poor venous access or needle-phobia).
4. Planned or expected major surgical procedure during the clinical study.
5. Patient is unwilling to refrain from using prohibited medications during the clinical study.
6. Currently participating or participated in any other clinical study of a drug or device, within the past 4 months before screening, or is in an exclusion period (if verifiable) from a previous study.

   Note: patients who have participated in Cohort 1 of this study may be enrolled to Cohort 2 after a minimum of 4 weeks from last KM-001 dose.
7. Cutaneous infection or another active underlying skin condition, regardless of location.
8. Cutaneous infection of the area to be applied with KM-001, requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals, or any topical treatments during and/or up-to 2 weeks before screening.
9. Pregnant or breastfeeding.
10. Failure to convince the investigator of fitness to participate in the study for any other reason.
11. Having received any of the prohibited treatments in Table 4 (Section 5.8) within the specified timeframe before baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Safety endpoint will be assessed through collection and analysis of adverse events | up to 91 days for arm 1 and 126 days for arm 2
  Incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs) grouped by body system will assessed.
Safety endpoint-will be assessed through collection and analysis of blood laboratory tests. | up to 91 days for arm 1 and 126 days for arm 2
  Data management team will assess and review the lab test results (blood), assessment will be compared to the normal range. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint-will be assessed through collection and analysis of urine laboratory tes | up to 91 days for arm 1 and 126 days for arm 2
  Data management team will assess and review the lab test results (urine), assessment will be compared to the normal range. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint-Vital signs- Heart rate | up to 91 days for arm 1 and 126 days for arm 2
  Vital signs (resting heart rate, systolic and diastolic blood pressure) will be assesed and the changes from the baseline.
  units: BPM (beats per minute) Data management team will assess and review the vital signs. The category of the assessments will be compared to the normal ranges. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint-Vital signs- Blood Pressure | up to 91 days for arm 1 and 126 days for arm 2
  Vital signs (resting heart rate, systolic and diastolic blood pressure) will be assesed and the changes from the baseline.
  units:blood pressure [mm Hg]. Data management team will assess and review the vital signs. The category of the assessments will be compared to the normal ranges. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoint-ECG | up to 91 days for arm 1 and 126 days for arm 2
  A 12-lead, resting, digital ECG will be taken for each participant at Screening and on Days 42 and 84, after the patient has been supine for at least 5 min. At minimum, the following ECG parameters will be recorded: heart rate (HR), PR, QT and QRS intervals and QTC. Resting ECG parameter and changes from baseline will be assesed
Safety endpoint- Lesion Assessment | up to 91 days for arm 1 and 126 days for arm 2
  Lesions severity will be assessed using the Investigator's Global Assessment (IGA) scale, which is a 5-point scale (from 0 ="no disease" to 4="severe disease").

SECONDARY OUTCOMES:
Pharmacokinetic profile of the study drug- maximal concentartion- Cmax | up to 91 days for arm 1 and 126 days for arm 2
  CMAX measurement (mg/ml)
Pharmacokinetic profile of the study drug- Time to reach Cmax - Tmax | up to 91 days for arm 1 and 126 days for arm 2
  Tmax measurement (h)
Pharmacokinetic profile of the study drug- AUC | up to 91 days for arm 1 and 126 days for arm 2
  AUC measurement (mg*h/L)
Efficacy endpoint- Investigator's Global Impression (IGA) score. | up to 84 days for arm 1 and 112 days for arm 2
  Effect of the treatment on target lesions, as assessed by change from baseline to each post baseline in-clinic visit in Investigator's Global Impression (IGA) score.
  Lesions severity will be assessed using the Investigator's Global Assessment (IGA) scale, which is a 5-point scale (from 0 ="no disease" to 4="severe disease") based on Simpson et al. 2020, IGA for atopic dermatitis (see Table 4; Simpson et al. 2020).
  The IGA score is selected using the descriptors below that best describe the overall appearance of the lesions at a given timepoint. It is not necessary that all characteristics under morphological description are present. Excoriations should not be considered when assessing disease severity.
Efficacy endpoint- Patient Global Impression of Change scoring | up to 84 days for arm 1 and 112 days for arm 2
  Mean score of Patient Global Impression of Change (PGI-C) on each post baseline in-clinic visit.
  The PGI-C will be evaluated using a 7-point scale from 1 (very much improved) to 7 (very much worse) answering the question Since the start of the trial, my overall status has.
Efficacy endpoint- Patient Global Impression of Severity scoring | up to 84 days for arm 1 and 112 days for arm 2
  Mean change from baseline in Patient Global Impression of Severity (PGI-S) to each post baseline in-clinic visit.
  The PGI-S will be evaluated using a 5-point scale from 1 (none) to 5 (very severe) answering the question Please rate the severity of your disease right now.
Efficacy endpoint- Visual Analogue Scale | up to 84 days for arm 1 and 112 days for arm 2
  Mean change from baseline in pain, assessed by Visual Analogue Scale (VAS) score, to each post baseline in-clinic visit.
  The following parameter will be evaluated on a VAS from 0 (no pain) to 100 (severe intolerable pain) based on the question: "How was your worst pain intensity in the past 24 hours?"

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Rabin Medical Center (Beilinson, Hasharon), Petah Tikva
  - Sourasky Medical Center - Ichilov Hospital, Tel Aviv

IPD SHARING:
Plan to Share IPD: No